CLINICAL TRIAL: NCT06520215
Title: Correlation Hand Grip Strength and Walking Distance in Elderly
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: IKFR-202407.01
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Coronary Revascularization

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly patient post coronary revascularization assessed hand grip strength and changes in six minute walking distance

DETAILED DESCRIPTION:
Coronary artery disease causes muscle dysfunction which leads to decreased muscle fitness due to reduced cardiac output, resulting in reduced oxygen uptake from the blood, and further decreases functional capacity or maximum oxygen uptake. The elderly population is an age group at risk of developing coronary artery disease. Handgrip strength s a good predictor for assessing overall muscle fitness, where handgrip strength assessment with a dynamometer is one method of determining muscle fitness, one of the factors affecting cardiorespiratory fitness, which can be assessed by the 6-minute walk test. This study wants to determine the correlation between handgrip strength and changes in 6-minute walk test after undergoing phase 2 cardiac rehabilitation in the elderly after coronary revascularization and this study also wants to know the predictive value using the parameters studied.

ELIGIBILITY:
Inclusion Criteria:

* Post coronary revascularization
* MMSE >= 26 BMI 18.5-25

Exclusion Criteria:

* Comorbid cardiovascular, lung, kidney and metabolic disease
* Frailty Syndrome

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient above 60 years
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Correlation Between Hand Grip Strength and Walking Distance in Elderly Patients | 6 weeks
  Elderly patient post coronary revascularization assessed hand grip strength (measured with hand dynamometer) and changes in six minute walking distance (measured in meter)

CONTACTS AND LOCATIONS:
Overall Officials: Irma Ruslina Defi, Principal Investigator — Padjadjaran University
Locations (1):
- Hasan Sadikin Hospital, Bandung, West Java, Indonesia